CLINICAL TRIAL: NCT03909971
Title: A PHASE 2, MULTI-CENTER, OPEN-LABEL, DUAL-COHORT STUDY TO EVALUATE THE EFFICACY AND SAFETY OF LORLATINIB (PF-06463922) MONOTHERAPY IN ALK INHIBITOR-TREATED LOCALLY ADVANCED OR METASTATIC ALK-POSITIVE NON-SMALL CELL LUNG CANCER PATIENTS IN CHINA
Brief Title: A Study of Lorlatinib in ALK Inhibitor-Treated ALK-Positive NSCLC in China
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B7461024; NCT03909971 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2019-02-05; First posted 2019-04-10 (Actual); Results first posted 2021-10-26 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: ALK positive; ALK inhibitor-treated; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lorlatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lorlatinib (Experimental): Lorlatinib single agent, 100 mg (4 x 25 mg) oral tables, QD, continuously
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — ALK inhibitor-treated ALK-positive NSCL treatment
  Other Names: PF-06463922

SUMMARY:
A Phase 2, multi center, open label, dual cohort study to evaluate the efficacy and safety of lorlatinib (PF 06463922) monotherapy in ALK inhibitor treated locally advanced or metastatic ALK positive non small cell lung cancer patients in China

DETAILED DESCRIPTION:
This is a Phase 2, China only, multi center, open label, dual cohort study, in ALK positive locally advanced or metastatic NSCLC patients will be enrolled to receive lorlatinib monotherapy.

* (in Cohort 1) Disease progression after crizotinib as the only ALK inhibitor.
* (in Cohort 2) Disease progression after one ALK inhibitor other than crizotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of histologically or cytologically confirmed diagnosis of locally advanced or metastatic ALK positive NSCLC where ALK status has been previously established by the Ventana ALK (D5F3) CDx Assay (Roche Diagnostics), the Vysis ALK Break Apart FISH Probe Kit (Abbott Molecular), or the EML4 ALK Fusion Gene Detection Kit (AmoyDx).
2. Subject should have:

   1. (in Cohort 1) Disease progression after crizotinib as the only ALK inhibitor;
   2. (in Cohort 2) Disease progression after one ALK inhibitor other than crizotinib, with or without prior crizotinib.
3. Prior treatment with an ALK inhibitor must have completed 5 half lives prior to study entry.
4. All Subjects must have at least 1 measurable extracranial target lesion according to RECIST v1.1 that has not been previously irradiated. CNS metastases are allowed if:

   1. Asymptomatic: either not currently requiring corticosteroid treatment, or on a stable or decreasing dose of 10 mg QD prednisone or equivalent; or
   2. Previously diagnosed and treatment has been completed with full recovery from the acute effects of radiation therapy or surgery prior to enrollment, and if corticosteroid treatment for these metastases has been withdrawn for at least 4 weeks with neurological stability.
5. Eastern Cooperative Oncology Group performance status (ECOG PS) 0, 1, or 2.
6. Age 18 years (or 20 years as required by local regulation).
7. Adequate bone marrow functions:

   1. Absolute Neutrophil Count (ANC) 1,500/mm3 or 1.5 x 109/L;
   2. Platelets 100,000/mm3 or 100 x 109/L;
   3. Hemoglobin 9 g/dL.
8. Adequate pancreatic function:

   1. Serum total amylase 1.5 x upper limit of normal (ULN);*
   2. Serum lipase 1.5 x ULN. *if total amylase >1.5 x ULN, but pancreatic amylase is within the ULN, then subject may be enrolled.
9. Adequate renal function:

   a. Serum creatinine 1.5 x ULN or estimated creatinine clearance 60 mL/min as calculated using the method standard for the institution.
10. Adequate liver function:

    1. Total serum bilirubin 1.5 x ULN;
    2. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) 2.5 x ULN (5.0 x ULN in case of liver metastases).
11. Acute effects of prior radiotherapy and chemotherapy resolved to baseline severity or to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 except for AEs that in the investigator's judgment do not constitute a safety risk for the subject.
12. Serum or urine pregnancy test (for females of childbearing potential) negative at screening. Female subjects of non childbearing potential must meet at least 1 of the following criteria:

    1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause (which may be confirmed with a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state if appropriate;
    2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
    3. Have medically confirmed ovarian failure. All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential.
13. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
14. Willing and able to comply with the study scheduled visits, treatment plans, laboratory tests, and other procedures.

Exclusion Criteria:

Subjects with any of the following characteristics/conditions will not be included in the study:

1. More than 1 prior chemotherapy regimen prior to enrollment in advanced/metastatic setting.

   If disease recurred/relapsed within the adjuvant chemotherapy treatment or <=6 months after the completion of the adjuvant chemotherapy, then the adjuvant chemotherapy is considered as the first line systemic chemotherapy to the disease.
2. Systemic anti cancer therapy completed within a minimum of 5 half lives of study enrollment.
3. Prior therapy with an antibody or drug specifically targeting T cell co stimulation or immune checkpoint pathways, including, but not limited to, anti programmed cell death protein 1 (anti PD 1), anti programmed cell death protein ligand 1 (anti PD L1), anti PD L2, anti cluster of differentiation 137 (anti CD137), or anti cytotoxic T lymphocyte associated antigen 4 (anti CTLA 4) antibody.
4. Known epidermal growth factor receptor (EGFR) activating mutations; known prior therapy with EGFR TKI(s) (the prior treatment with brigatinib is allowed as an ALK TKI).
5. Major surgery within 4 weeks prior to enrollment. Minor surgical procedures (eg, port insertion) are not excluded, but sufficient time should have passed for adequate wound healing.
6. Radiation therapy within 2 weeks prior to enrollment. Palliative radiation must have been completed at least 48 hours prior to enrollment. Stereotactic or partial brain irradiation must have completed at least 2 weeks prior to enrollment. Whole brain irradiation must have completed at least 4 weeks prior to enrollment.
7. Spinal cord compression unless the subject has good pain control attained through therapy, and there is complete recovery of neurological function for the 4 weeks prior to enrollment.
8. Gastrointestinal abnormalities, including inability to take oral medication; requirement for intravenous alimentation; prior surgical procedures affecting absorption including total gastric resection or lap band; active inflammatory gastrointestinal disease, chronic diarrhea, symptomatic diverticular disease; treatment for active peptic ulcer disease in the past 6 months; malabsorption syndromes.
9. Known prior or suspected severe hypersensitivity to lorlatinib or any component in the formulation; known prior therapy with lorlatinib.
10. Active and clinically significant bacterial, fungal, or viral infection including hepatitis B virus (HBV), hepatitis C virus (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness.
11. Clinically significant cardiovascular disease (both arterial and venous) and non vascular cardiac conditions, (active or within 3 months prior to enrollment, which may include, but not are limited to:

    * Arterial disease such as cerebral vascular accident/stroke (including transient ischemic attack -TIA), myocardial infarction, unstable angina;
    * Venous diseases such as cerebral venous thrombosis, symptomatic pulmonary embolism;
    * Nonvascular cardiac disease such as congestive heart failure (New York Heart Association Classification Class ≥ II), second degree or third degree atrioventricular block (unless paced) or any AV block with PR interval >220 msec; or
    * Ongoing cardiac dysrhythmias of CTCAE Grade ≥2, uncontrolled atrial fibrillation of any grade, bradycardia defined as <50 bpm (unless subject is otherwise healthy such as long distance runners, etc.), machine read electrocardiogram (ECG) with QTc >470 msec, or congenital long QT syndrome.
12. Subject with predisposing characteristics for acute pancreatitis according to investigator judgment, including but not limited to uncontrolled hyperglycemia, current gallstone disease, in the last month prior to enrollment.
13. History of extensive, disseminated, bilateral or presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis and pulmonary fibrosis.
14. Evidence of active malignancy (other than NSCLC, non melanoma skin cancer, or localized and presumed cured prostate cancer or any in situ cancer which does not currently require treatment) within the last 3 years prior to enrollment.
15. Concurrent use of any of the following food or drugs (consult the sponsor if in doubt whether a food or a drug falls into any of the above categories) within 12 days prior to the first dose of administration of lorlatinib:

    1. Known strong CYP3A inhibitors (eg, strong CYP3A inhibitors: grapefruit juice or grapefruit/grapefruit related citrus fruits [eg, Seville oranges, pomelos], boceprevir, cobicistat, conivaptan, itraconazole, ketoconazole, posaconazole, ritonavir alone and with danoprevir or elvitegravir or indinavir or lopinavir or paritaprevir or ombitasvir or dasabuvir or saquinavir or tipranavir, telaprevir, troleandomycin, and voriconazole). The topical use of these medications (if applicable), such as 2% ketoconazole cream, is allowed;
    2. Known CYP3A substrates with narrow therapeutic index, such as astemizole*, terfenadine*, cisapride*, pimozide, quinidine, tacrolimus, cyclosporine, sirolimus, alfentanil, fentanyl (including transdermal patch) or ergot alkaloids (ergotamine, dihydroergotamine) (*withdrawn from US market);
    3. Known strong CYP3A inducers (eg, carbamazepine, enzalutamide, mitotane, phenytoin, rifampin, St. John's Wort);
    4. Known P glycoprotein (P gp) substrates with a narrow therapeutic index (eg, digoxin).
16. Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator and/or the sponsor, would make the subject inappropriate for entry into this study.
17. Subject who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
18. Participation in other studies involving investigational drug(s) within 2 weeks prior to study entry and/or during study participation.
19. Pregnant female participants; breastfeeding female participants; fertile male participants and female participants of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 97 days if male or 35 days if female, after the last dose of investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-04-28 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2024-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- China (21):
  - Gaoxin Hospital of The First Affilated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Province Oncology Hospital, Fuzhou, Fujian
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hunan Provincial Tumor Hospital/Division of Oncology, Changsha, Hunan
  - The first hospital of jilin university, Changchun, Jilin
  - Jilin Provincial Cancer Hospital, Changchun, Jilin
  - Tangdu Hospital of Fourth Military Medical University, Xi’an, Shanxi
  - Sichuan Province Cancer Hospital/Department of Pulmonary Tumor, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Cancer center, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of College of Medicine of Zhejiang University, Center for Oncology, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Fifth Medical Center of PLA General Hospital, Beijing
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - General Hospital of Eastern Theater Command, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Lu S, Zhou Q, Liu X, Du Y, Fan Y, Cheng Y, He S, Zhao H, Li H, Wu YL. Updated Efficacy and Safety of Lorlatinib in a Phase 2 Study in Chinese Patients With Previously Treated Advanced ALK-Positive Non-small Cell Lung Cancer. Clin Lung Cancer. 2024 Nov;25(7):e295-e303.e4. doi: 10.1016/j.cllc.2024.04.017. Epub 2024 Apr 30. PMID 38879393
- [Derived] Niu R, Zhang Y, Pang J, Zhou Q, Lei Y, Du Y. Effective treatment of advanced lung adenocarcinoma with paraneoplastic leukemoid reaction with Lorlatinib: a case report. Front Oncol. 2024 Jan 26;14:1341233. doi: 10.3389/fonc.2024.1341233. eCollection 2024. PMID 38344203
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461024

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled 109 participants, with 67 in Cohort 1 and 42 in Cohort 2.
Groups:
- Cohort 1: Participants whose disease had progressed after crizotinib as the only anaplastic lymphoma kinase (ALK) inhibitor were enrolled in Cohort 1 to receive lorlatinib 100 mg orally once daily (QD) continuously until confirmed disease progression by Independent Central Radiology (ICR) (unless clinical benefit is still achievable), participant refusal, participant lost to follow-up, unacceptable toxicity, or the study is terminated by the sponsor, whichever comes first. Each cycle duration was 21 days.
- Cohort 2: Participants whose disease had progressed after one ALK inhibitor treatment other than crizotinib, with or without prior crizotinib were enrolled in Cohort 2 to receive lorlatinib100 mg QD continuously until confirmed disease progression by ICR (unless clinical benefit is still achievable), participant refusal, participant lost to follow-up, unacceptable toxicity, or the study is terminated by the sponsor, whichever comes first. Each cycle duration was 21 days.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 67 | 42
Completed | 0 | 0
Not Completed | 67 | 42
Not completed — Participant transition to rollover study | 26 | 9
Not completed — Global Deterioration of Health Status | 2 | 2
Not completed — Progressive Disease | 28 | 21
Not completed — Death | 6 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Participant was unwilling to come to site visit | 0 | 1
Not completed — No longer benefit from Lorlatinib | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Participants whose disease had progressed after crizotinib as the only ALK inhibitor were enrolled in Cohort 1 to receive lorlatinib 100 mg orally QD continuously until confirmed disease progression by ICR (unless clinical benefit is still achievable), participant refusal, participant lost to follow-up, unacceptable toxicity, or the study is terminated by the sponsor, whichever comes first. Each cycle duration was 21 days.
- Cohort 2: Participants whose disease had progressed after one ALK inhibitor treatment other than crizotinib, with or without prior crizotinib were enrolled in Cohort 2 to receive lorlatinib 100 mg QD continuously until confirmed disease progression by ICR (unless clinical benefit is still achievable), participant refusal, participant lost to follow-up, unacceptable toxicity, or the study is terminated by the sponsor, whichever comes first. Each cycle duration was 21 days.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 67 | 42 | 109
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.4 (10.85) | 52.1 (13.36) | 51.0 (11.84)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 35 | 96
  >65 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 23 | 56
  Male | 34 | 19 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian: Chinese | 67 | 42 | 109

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (Cohort 1)
Description: Objective response rate (ORR) was defined as the percentage of participants with a best overall confirmed response of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1 relative to the total participants in the analysis population. CR was defined as the disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeter (mm). PR was defined as a greater than equal to (>=) 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. Independent Central Radiology (ICR) was used for disease progression assessment.
Time Frame: From Cycle 1 Day 1 to documented progression of disease by ICR (up to 67 weeks)
Population: The analysis population included all enrolled participants who received at least 1 dose of lorlatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 67
Percentage of participants | 70.1 [57.7 to 80.7]
Statistical Analysis 1: Comparison: Cohort 1; Test type: Superiority; p < 0.0001, Fisher Exact

2. Other Pre Specified Outcome: Percentage of Participants With Objective Response (Cohort 1)-Final Analysis
Description: ORR was defined as the percentage of participants with a best overall confirmed response of CR or PR according to RECIST version 1.1 relative to the total participants in the analysis population. CR was defined as the disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. ICR was used for disease progression assessment.
Time Frame: From first dose (Cycle 1 Day 1) to documented disease progression by ICR (up to 271 weeks of treatment exposure)
Population: The safety analysis population included all enrolled participants who received at least 1 dose of lorlatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 67
Percentage of participants | 79.1 [67.4 to 88.1]

3. Secondary Outcome: Percentage of Participants With Objective Response (Cohort 2)
Description: as for outcome 2
Time Frame: From Cycle 1 Day 1 to documented progression of disease by ICR (up to 67 weeks)
Population: The analysis population included all enrolled participants who received at least 1 dose of loratinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2
Number analyzed (Participants) | 42
Percentage of participants | 47.6 [32.0 to 63.6]

4. Secondary Outcome: Progression-Free Survival (PFS) Based on ICR Assessment
Description: PFS was defined as the time from first dose to first documentation of objective disease progression (PD) or to death due to any cause, whichever came first. PD: at least a >=20 percent (%) increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. For non-target lesions, PD was defined as unequivocal progression of existing non-target lesions, or the appearance of >=1 new lesion. Participants without documentation of PD, or death at the time of analysis were censored at the date of the last tumor assessment. Analysis was performed using Kaplan Meier method. ICR was used for disease progression assessment.
Time Frame: From first dose (Cycle 1 Day 1) to documented PD by ICR, death due to any cause or date of censoring, whichever occurred first (up to 271 weeks of treatment exposure)
Population: The safety analysis population included all enrolled participants who received at least 1 dose of lorlatinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 67 | 42
Months | 26.3 [16.6 to NA] — Upper limit of 95% confidence interval (CI) could not be estimated due to insufficient number of participants with events. | 5.6 [2.9 to 12.4]

5. Secondary Outcome: Progression-Free Survival Based on Investigator Assessment
Description: PFS was defined as the time from first dose to first documentation of objective PD or to death due to any cause, whichever came first. PD: at least a >=20 % increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. For non-target lesions, PD was defined as unequivocal progression of existing non-target lesions, or the appearance of >=1 new lesion. Participants without documentation of PD, or death at the time of analysis were censored at the date of the last tumor assessment. Analysis was performed using Kaplan Meier method. Investigator assessment was used for disease progression assessment.
Time Frame: From first dose (Cycle 1 Day 1) to documented progression of disease by investigator, death due to any cause or date of censoring, whichever occurred first (up to 271 weeks of treatment exposure)
Population: The safety analysis population included all enrolled participants who received at least 1 dose of lorlatinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 67 | 42
Months | 26.3 [15.2 to 52.4] | 6.9 [4.2 to 13.7]

6. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from first dose to the date of death due to any cause. Analysis was performed using Kaplan Meier method.
Time Frame: From first dose (Cycle 1 Day 1) to date of death due to any cause (up to 271 weeks of treatment exposure)
Population: The safety analysis population included all enrolled participants who received at least 1 dose of lorlatinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 67 | 42
Months | NA [42.7 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 21.9 [11.9 to 44.1]

7. Secondary Outcome: Percentage of Participants With Intracranial Objective Response (IC-OR) Based on ICR Assessment
Description: IC-OR: percentage of participants with a best overall confirmed intracranial response of CR or PR according to RECIST version 1.1 relative to total participants in the analysis population but limited to intra cranial lesions only in participants with central nervous system metastases. CR was defined as the disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as a >= 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. 95% CI was based on Clopper-Pearson method.
Time Frame: From first dose (Cycle 1 Day 1) to documented PD by ICR (up to 271 weeks of treatment exposure)
Population: The safety analysis population included all enrolled participants who received at least 1 dose of lorlatinib. Here, 'Overall Number of Participants Analyzed' signifies participants for whom the brain lesions were chosen as RECIST target or non-target lesions at baseline and who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 37 | 22
Percentage of participants | 83.8 [68.0 to 93.8] | 50.0 [28.2 to 71.8]

8. Secondary Outcome: Percentage of Participants With Intracranial Objective Response Based on Investigator Assessment
Description: as for outcome 7
Time Frame: From first dose (Cycle 1 Day 1) to documented progression of disease by investigator (up to 271 weeks of treatment exposure)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 41 | 24
Percentage of participants | 63.4 [46.9 to 77.9] | 33.3 [15.6 to 55.3]

9. Secondary Outcome: Duration of Response (DOR) Based on ICR Assessment
Description: DOR: time from first documentation of CR or PR to first documentation of PD or death due to any cause, whichever occurred first. CR: disappearance of all target lesions and non-target lesions. Any pathological lymph nodes must have reduction in short axis to <10mm. PR:>=30% decrease in sum of longest dimensions of target lesions taking as a reference baseline sum longest dimensions. PD:>=20 % increase in sum of longest dimensions of target lesions taking as a reference smallest sum of longest dimensions recorded since treatment started, or the appearance of one or more new lesions. In addition to relative increase of 20% sum must also demonstrate an absolute increase of at least 5 mm and for non-target lesions PD: unequivocal progression of existing non-target lesions or the appearance of >=1 new lesion. Participants without documentation of PD, or death at time of analysis were censored at date of last tumor assessment. Analysis was performed using Kaplan Meier method.
Time Frame: From first documentation of CR or PR to documented progression of disease by ICR, death due to any cause or date of censoring, whichever occurred first (up to 271 weeks of treatment exposure)
Population: The safety analysis population included all enrolled participants who received at least 1 dose of lorlatinib. Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 53 | 20
Months | 31.7 [18.0 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 10.4 [2.9 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events.

10. Secondary Outcome: DOR Based on Investigator Assessment
Description: as for outcome 9
Time Frame: From first documentation of CR or PR to documented PD by investigator, death due to any cause or date of censoring, whichever occurred first (up to 271 weeks of treatment exposure
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 47 | 17
Months | 20.9 [12.4 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 20.8 [5.6 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events.

11. Secondary Outcome: Duration of Intracranial Response Based on ICR Assessment
Description: Duration of intracranial response: time from first documentation of CR or PR considering only lesions having disease site=brain to first documentation of PD or death due to any cause, whichever occurred first, participants who had at least 1 intracranial lesion.CR: disappearance of all target and non-target lesions. Any pathological lymph nodes must have reduction in <10mm.PR:>=30% decrease in the sum of the longest dimensions of target lesions taking reference the baseline sum longest dimension. PD:>=20% increase in sum of longest dimensions of target lesion, or appearance of one or more new lesion. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5mm and for non-target lesion PD: unequivocal progression of existing non-target lesion, or the appearance of >=1 new lesion. Participants without documentation of PD, or death at the time of analysis were censored at the date of the last tumor assessment. Kaplan Meier method was used.
Time Frame: as for outcome 9
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 31 | 11
Months | NA [30.6 to NA] — Median and upper limit of 95% CI were not estimable due to insufficient number of participants with events. | NA [5.6 to NA] — Median and upper limit of 95% CI were not estimable due to insufficient number of participants with events.

12. Secondary Outcome: Duration of Intracranial Response Based on Investigator Assessment
Description: Duration of intracranial response: time from first documentation of CR or PR considering only lesions having disease site=brain to first documentation of PD or death due to any cause, whichever occurred first, participants who had at least 1 intracranial lesion.CR: disappearance of all target and non-target lesions. Any pathological lymph nodes must have reduction in <10mm.PR:>=30% decrease in the sum of the longest dimensions of target lesions taking reference the baseline sum longest dimension. PD:>=20% increase in sum of longest dimensions of target lesion or appearance of one or more new lesion. In addition to relative increase of 20% sum must also demonstrate an absolute increase of at least 5mm and for non-target lesion PD: unequivocal progression of existing non-target lesion, or the appearance of >=1 new lesion. Participants without documentation of PD, or death at the time of analysis were censored at the date of the last tumor assessment. Kaplan Meier method was used.
Time Frame: From first documentation of CR or PR to documented progression of disease by investigator, death due to any cause or date of censoring, whichever occurred first (up to 271 weeks of treatment exposure)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 26 | 8
Months | NA [15.1 to NA] — Median and upper limit of 95% CI were not estimable due to insufficient number of participants with event. | NA [8.3 to NA] — Median and upper limit of 95% CI were not estimable due to insufficient number of participants with event.

13. Secondary Outcome: Time to Tumor Response Based on ICR Assessment
Description: Time to tumor response was defined as the time from first dose to first documentation of objective tumor response CR or PR. CR was defined as the disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From first dose (Cycle 1 Day 1) to first documented CR or PR (up to 271 weeks of treatment exposure)
Population: as for outcome 9
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 53 | 20
Months | 1.4 [1.2 to 17.9] | 1.4 [1.2 to 6.9]

14. Secondary Outcome: Time to Tumor Response Based on Investigator Assessment
Description: as for outcome 13
Time Frame: From first dose (Cycle 1 Day 1) to documented first CR or PR (up to 271 weeks of treatment exposure)
Population: as for outcome 9
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 47 | 17
Months | 1.4 [1.2 to 27.6] | 1.4 [1.2 to 17.9]

15. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE:any untoward medical occurrence in a study participant administered a product or medical device;event did not necessarily have a causal relationship with treatment or usage.Serious AE:any untoward medical occurrence at any dose resulted in death;life-threatening;required inpatient or prolongation of existing hospitalization;persistent or significant disability/incapacity; congenital anomaly/birth defect or that was considered to be an important event.AEs were graded by the National Cancer Institute Common Terminology Criteria AE(NCICTCAE)v4.03 where,Grade(G)1:mild AE;G2:moderate;G3:severe;G4:life-threatening consequences,urgent intervention indicated;G5:death related to AE. Focus of AE summaries was on treatment-emergent AE(TEAE).AE was considered TEAE if the event occurred during the on-treatment period.On-treatment:time from first dose of study treatment through end of study follow-up(i.e.,up to 28 days after last dose of treatment. Participant with G3or4 and5 AEs were reported.
Time Frame: From start of study treatment (Cycle 1 Day 1) up to 28 days after the last administration of the investigational product, up to approximately 275 weeks
Population: The safety analysis population included all enrolled participants who received at least 1 dose of lorlatinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 67 | 42
Participants
  All-causality TEAEs | 67 | 42
  Treatment-related TEAEs | 67 | 42
  All-causality serious AEs | 23 | 16
  Treatment-related serious AEs | 11 | 5
  All-causalities maximum Grade 3 or 4 AEs | 49 | 25
  Treatment-related Grade 3 or 4 AEs | 46 | 19
  All-causality Grade 5 AEs | 4 | 7
  Treatment-related Grade 5 AEs | 0 | 0

16. Secondary Outcome: Number of Participants With Central Nervous System-Related Adverse Events
Description: An AE was any untoward medical occurrence in a study participant administered a product or medical device; the event did not necessarily have a causal relationship with the treatment or usage. The central-nervous system-related AEs included AEs under the cluster terms of mood effects, cognitive effects, psychotic effects, and speech effects.
Time Frame: as for outcome 15
Population: The safety analysis population included all enrolled participants who received at least 1 dose of lorlatinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 67 | 42
Participants
  Cognitive Effects | 2 | 1
  Mood Effects | 1 | 2
  Speech Effects | 0 | 1
  Psychotic Effects | 1 | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities
Description: Laboratory tests included hematology, chemistry and lipids. Laboratory test results were graded according to NCI CTCAE version 4.03, where Grade 0: no AE, Grade 1 : mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. Shifts from Grade <=2 at baseline to Grade 3 or 4 post-baseline were considered clinically significant. Only categories with non-zero values were reported in this outcome measure.
Time Frame: as for outcome 15
Population: The safety analysis population included all enrolled participants who received at least 1 dose of Lorlatinib. Here, "Number Analyzed" signifies number of participants evaluable for each row.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 67 | 42
Participants
  Anemia: Grade 0 to Grade 3 or 4 | 3 | 0
  Anemia:Grade 1 to Grade 3 or 4 | 2 | 3
  Anemia:Grade 2 to Grade 3 or 4 | 1 | 1
  Lymphocyte count decreased Grade 0 to Grade 3 or 4 | 3 | 0
  Lymphocyte count decreased:Grade 1 to Grade 3 or 4 | 1 | 0
  Platelet count decreased: Grade 0 to Grade 3 or 4 | 2 | 1
  Alanine aminotransferase increased: Grade 0 to Grade 3 or 4 | 2 | 0
  Alanine aminotransferase increased:Grade 1 to Grade 3 or 4 | 2 | 0
  Alkaline phosphatase increased: Grade 0 to Grade 3 or 4 | 1 | 0
  Aspartate aminotransferase increased: Grade 0 to Grade 3 or 4 | 2 | 1
  Aspartate aminotransferase increased:Grade 1 to Grade 3 or 4 | 1 | 0
  Blood bilirubin increased: Grade 0 to Grade 3 or 4 | 1 | 0
  Blood bilirubin increased:Grade 1 to Grade 3 or 4 | 0 | 1
  CPK increased: Grade 0 to Grade 3 or 4: number analyzed (Participants) | 53 | 33
  CPK increased: Grade 0 to Grade 3 or 4 | 0 | 1
  CPK increased:Grade 2 to Grade 3 or 4: number analyzed (Participants) | 53 | 33
  CPK increased:Grade 2 to Grade 3 or 4 | 1 | 0
  Creatinine increased: Grade 0 to Grade 3 or 4 | 1 | 1
  GGT increased: Grade 0 to Grade 3 or 4 | 3 | 2
  GGT increased:Grade 1 to Grade 3 or 4 | 2 | 0
  Hypercalcemia: Grade 0 to Grade 3 or 4 | 0 | 1
  Hyperglycemia: Grade 0 to Grade 3 or 4 | 6 | 0
  Hyperglycemia:Grade 1 to Grade 3 or 4 | 1 | 1
  Hypermagnesemia: Grade 0 to Grade 3 or 4 | 7 | 1
  Hypocalcemia: Grade 0 to Grade 3 or 4 | 0 | 1
  Hypokalemia: Grade 0 to Grade 3 or 4 | 2 | 2
  Hypokalemia:Grade 2 to Grade 3 or 4 | 1 | 0
  Hyponatremia: Grade 0 to Grade 3 or 4 | 1 | 1
  Hyponatremia:Grade 1 to Grade 3 or 4 | 0 | 1
  Hypophosphatemia: Grade 0 to Grade 3 or 4 | 4 | 1
  Hypophosphatemia:Grade 1 to Grade 3 or 4 | 0 | 1
  Lipase increased: Grade 0 to Grade 3 or 4 | 5 | 2
  Lipase increased:Grade 1 to Grade 3 or 4 | 1 | 0
  Serum amylase increased: Grade 0 to Grade 3 or 4 | 1 | 1
  Cholesterol high: Grade 0 to Grade 3 or 4 | 12 | 1
  Cholesterol high:Grade 1 to Grade 3 or 4 | 6 | 3
  Cholesterol high:Grade 2 to Grade 3 or 4 | 1 | 0
  Hypertriglyceridemia: Grade 0 to Grade 3 or 4 | 19 | 3
  Hypertriglyceridemia:Grade 1 to Grade 3 or 4 | 9 | 6
  Hypertriglyceridemia:Grade 2 to Grade 3 or 4 | 3 | 1

18. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Pre-specified Criteria
Description: Vital signs evaluation included diastolic blood pressure (DBP), systolic blood pressure (SBP), pulse rate and weight. Blood pressure and pulse rate were recorded in sitting position after the participant had been sitting quietly for at least 5 minutes. The pre-specified criteria included: sitting SBP change >=40 millimeters of mercury (mmHg) increase, >=40 mmHg decrease; sitting DBP change >=20 mmHg increase, change >=20 mmHg decrease, or change >=60 mmHg increase; sitting pulse rate value <50 beats per minute (bpm), >120 bpm, change >=30 bpm increase, or change >=30 bpm decrease; weight 10% <= change <20% increase, change >=20% increase or change >=10% decrease. One participant can have more than one vital sign data meeting pre-specified criteria.
Time Frame: as for outcome 15
Population: The safety analysis population included all enrolled participants who received at least 1 dose of lorlatinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 67 | 42
Participants
  Sitting SBP change >=40 mmHg increase | 10 | 1
  Sitting SBP change >=40 mmHg decrease | 2 | 0
  Sitting DBP change >=20 mmHg increase | 26 | 10
  Sitting DBP change >=20 mmHg decrease | 12 | 7
  Sitting DBP change >=60 mmHg increase | 0 | 0
  Sitting pulse rate value <50 bpm | 0 | 0
  Sitting pulse rate value >120 bpm | 5 | 3
  Sitting pulse rate change >=30 mmHg increase | 18 | 5
  Sitting pulse rate change >=30 mmHg decrease | 5 | 7
  weight 10% <= change <20% kg increase | 43 | 22
  Weight change >=20% kg increase | 14 | 6
  Weight change >=10% kg decrease | 3 | 2

19. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-specified Criteria
Description: The QT intervals were corrected for heart rate (QTc) using standard correction factors (ie, QTcF [Fridericia's], QTcB [Bazett's], and possibly a study-specified factor, as appropriate). The pre-specified criteria included: PR interval change >= 50% and baseline <200 msec, change >=25% and baseline >=200 msec; QRS interval change >=50% and baseline <100 msec, change >=25% and baseline >=100 msec; QTcB values <=450 msec, 450 < Value <= 480 msec, 480 < Value <= 500 msec, value >500 msec, change <=30 msec, 30 < Change <= 60 msec, change >60 msec; QTcF value <=450 msec, 450 < Value <= 480 msec, 480 < Value <= 500 msec, Value > 500 msec, change <=30 msec, 30 < Change <=60 msec and change >60 msec. . One participant can have more than one ECG data meeting pre-specified criteria.
Time Frame: as for outcome 15
Population: The safety analysis population included all enrolled participants who received at least 1 dose of lorlatinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 67 | 42
Participants
  PR interval change >=50% and baseline <200 msec | 4 | 1
  PR interval change >=25% and baseline >=200 msec | 0 | 0
  QRS interval change >=50% and baseline<100 msec | 1 | 1
  QRS interval change >=25% and baseline >=100 msec | 2 | 0
  QTcB value <=450 msec | 27 | 27
  QTcB 450 < Value <= 480 msec | 26 | 9
  QTcB 480 < Value <= 500 msec | 5 | 3
  QTcB value >500 msec | 9 | 3
  QTcB change <=30 msec | 31 | 25
  QTcB 30 < Change <= 60 msec | 24 | 14
  QTcB change >60 msec | 12 | 3
  QTcF value <=450 msec | 49 | 35
  QTcF 450 < Value <= 480 msec | 13 | 6
  QTcF 480 < Value <= 500 msec | 1 | 1
  QTcF value >500 msec | 4 | 0
  QTcF change <=30 msec | 39 | 29
  QTcF 30 < Change <= 60 msec | 20 | 9
  QTcF change >60 msec | 8 | 4

20. Secondary Outcome: Number of Participants With Left Ventricular Ejection Fraction (LVEF) Meeting Pre-specified Criteria
Description: Echocardiogram or multigated acquisition scan were performed to monitor LVEF. Pre-specified criteria included shift from baseline normal to post-baseline below lower limit of normal (LLN) >=20-point decrease from baseline in LVEF% .
Time Frame: as for outcome 15
Population: The safety analysis population included all enrolled participants who received at least 1 dose of lorlatinib and who had at least 1 result of the LVEF value. Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 67 | 40
Participants
  LVEF change from baseline normal to post-baseline below LLN | 7 | 0
  LVEF >=20-point decrease from baseline | 3 | 0

21. Secondary Outcome: Cycle 1 Day 1 Maximum Plasma Concentration (Cmax)
Description: The loratinib Cmax was estimated using non-compartmental analysis.
Time Frame: At pre-dose, 0.5, 1, 2, 3, 4, 6 ,8, 9 and 24 hours on Cycle 1 Day 1
Population: The analysis population included all enrolled participants who received at least 1 dose of loratinib and had sufficient information to estimate at least 1 of the pharmacokinetic parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
nanogram per milliliter (ng/mL) | 1004 (42) | 1074 (58)

22. Secondary Outcome: Cycle 1 Day 1 Time to Cmax (Tmax)
Description: The loratinib Tmax was estimated using non-compartmental analysis.
Time Frame: At pre-dose, 0.5, 1, 2, 3, 4, 6 ,8, 9 and 24 hours on Cycle 1 Day 1
Population: as for outcome 21
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
hour | 1.02 [0.500 to 3.12] | 1.45 [0.483 to 4.00]

23. Secondary Outcome: Cycle 1 Day 1 Area Under the Plasma Concentration Versus Time Profile Within A Dose Interval (AUCtau)
Description: The loratinib AUCtau was estimated using non-compartmental analysis.
Time Frame: At pre-dose, 0.5, 1, 2, 3, 4, 6 ,8, 9 and 24 hours on Cycle 1 Day 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng.hr/mL)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
nanogram*hour per milliliter (ng.hr/mL) | 7310 (17) | 7778 (39)

24. Secondary Outcome: Steady-State Cmax
Description: The loratinib Cmax was estimated using non-compartmental analysis. Steady-state was reached on Cycle 1 Day 15.
Time Frame: At Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, and 24 hours on Day 15 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
ng/mL | 643.9 (50) | 795.9 (40)

25. Secondary Outcome: Steady-State Tmax
Description: The loratinib Tmax was estimated using non-compartmental analysis. Steady-state was reached on Cycle 1 Day 15.
Time Frame: At Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, and 24 hours on Day 15 of Cycle 1
Population: as for outcome 21
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
hour | 1.53 [0.533 to 3.03] | 1.88 [0.500 to 8.02]

26. Secondary Outcome: Steady-State AUCtau
Description: The loratinib AUCtau was estimated using non-compartmental analysis. Steady-state was reached on Cycle 1 Day 15.
Time Frame: At Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, and 24 hours on Day 15 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
ng*hr/mL | 5388 (37) | 6801 (40)

27. Secondary Outcome: Apparent Clearance (CL/F)
Description: The loratinib CL/F was estimated using non-compartmental analysis. Steady-state was reached on Cycle 1 Day 15.
Time Frame: At Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, and 24 hours on Day 15 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Liter per hour (L/hr) | 18.55 (37) | 14.71 (40)

28. Secondary Outcome: Observed Accumulation Ratio (Rac)
Description: The loratinib Rac was estimated using non-compartmental analysis. Steady-state was reached on Cycle 1 Day 15.
Time Frame: At Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, and 24 hours on Day 15 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Ratio | 0.7371 (47) | 0.9578 (33)

ADVERSE EVENTS:
Time Frame: From start of study treatment (Cycle 1 Day 1) up to 28 days after the last administration of the investigational product, up to approximately 275 weeks
Description: The same event may appear as both non-SAE and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. AE reporting, including suspected unexpected serious adverse reactions, was carried out in accordance with applicable local regulations.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 28/67 | 26/42
Serious Adverse Events (participants affected / at risk) | 23/67 | 16/42
Other Adverse Events (participants affected / at risk) | 67/67 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=67) | Cohort 2 (N=42)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Pericarditis constrictive (Cardiac disorders) | 1 | 0
Death (General disorders) | 0 | 1
Disease progression (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Sudden death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 5
Post procedural infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=67) | Cohort 2 (N=42)
Anaemia (Blood and lymphatic system disorders) | 31 | 15
Atrioventricular block first degree (Cardiac disorders) | 4 | 3
Sinus bradycardia (Cardiac disorders) | 6 | 5
Sinus tachycardia (Cardiac disorders) | 8 | 3
Ventricular extrasystoles (Cardiac disorders) | 1 | 4
Vision blurred (Eye disorders) | 6 | 1
Vomiting (Gastrointestinal disorders) | 4 | 3
Oedema peripheral (General disorders) | 14 | 9
Pain (General disorders) | 5 | 2
Peripheral swelling (General disorders) | 8 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 0
Hepatic steatosis (Hepatobiliary disorders) | 4 | 0
Alanine aminotransferase increased (Investigations) | 38 | 19
Albumin urine present (Investigations) | 2 | 3
Amylase increased (Investigations) | 12 | 4
Aspartate aminotransferase increased (Investigations) | 40 | 18
Blood alkaline phosphatase increased (Investigations) | 7 | 9
Blood cholesterol increased (Investigations) | 29 | 14
Blood creatinine increased (Investigations) | 12 | 6
Blood glucose increased (Investigations) | 6 | 4
Blood lactate dehydrogenase increased (Investigations) | 5 | 3
Blood triglycerides increased (Investigations) | 15 | 5
Blood urea increased (Investigations) | 6 | 3
Electrocardiogram QT prolonged (Investigations) | 20 | 9
Gamma-glutamyltransferase increased (Investigations) | 28 | 12
Haemoglobin decreased (Investigations) | 3 | 4
High density lipoprotein increased (Investigations) | 6 | 4
Lipase increased (Investigations) | 12 | 6
Low density lipoprotein increased (Investigations) | 13 | 10
Neutrophil count decreased (Investigations) | 12 | 3
Platelet count decreased (Investigations) | 14 | 3
Weight increased (Investigations) | 49 | 19
White blood cell count decreased (Investigations) | 7 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 41 | 29
Hyperglycaemia (Metabolism and nutrition disorders) | 31 | 6
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 60 | 32
Hyperuricaemia (Metabolism and nutrition disorders) | 17 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 3
Hypoaesthesia (Nervous system disorders) | 11 | 3
Haematuria (Renal and urinary disorders) | 8 | 4
Proteinuria (Renal and urinary disorders) | 7 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 0
Hypertension (Vascular disorders) | 13 | 5
Arrhythmia (Cardiac disorders) | 4 | 0
Left ventricular dysfunction (Cardiac disorders) | 4 | 0
Pericardial effusion (Cardiac disorders) | 6 | 3
Supraventricular extrasystoles (Cardiac disorders) | 3 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Chest discomfort (General disorders) | 5 | 1
Fatigue (General disorders) | 4 | 0
COVID-19 (Infections and infestations) | 5 | 3
Pneumonia (Infections and infestations) | 7 | 3
Sinusitis (Infections and infestations) | 4 | 0
Suspected COVID-19 (Infections and infestations) | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 2
Blood albumin decreased (Investigations) | 2 | 5
Blood bilirubin increased (Investigations) | 4 | 1
Blood creatine phosphokinase increased (Investigations) | 13 | 6
Blood phosphorus decreased (Investigations) | 1 | 3
Blood pressure increased (Investigations) | 2 | 5
Blood uric acid increased (Investigations) | 3 | 4
Lymphocyte count decreased (Investigations) | 2 | 4
SARS-CoV-2 test positive (Investigations) | 9 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 4 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Dizziness (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 4 | 1
Paraesthesia (Nervous system disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0
Pyrexia (General disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclosure previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT03909971/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT03909971/SAP_001.pdf